CLINICAL TRIAL: NCT05659212
Title: A Comparative Randomized Study Between Dexmedetomidine, Magnesium Sulphate and Lidocaine on the Pressor Response to Laryngoscopic Intubation for Laparoscopic Gynecological Surgery
Brief Title: Block Pressor Response to Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Assistant professor of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM 11 2022
Record Dates: First submitted 2022-11-25; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Intubation Complication
MeSH Terms: interventions — Dexmedetomidine; Magnesium Sulfate; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group D (Active Comparator): Patients will receive IV dexmedetomidine 0.5 μg /kg diluted up to 10 ml with normal saline infused over 10 min before induction of anesthesia, and 10 ml of normal saline immediately before induction of anesthesia.
  Interventions: Drug: Dexmedetomidine
- Group M (Active Comparator): Patients will receive IV magnesium sulphate 50 mg/kg diluted up to 10 ml with normal saline infused slowly over 10 min before induction of anesthesia, and 10 ml of normal saline immediately before induction of anesthesia.
  Interventions: Drug: Magnesium sulphate
- Group L (Placebo Comparator): Patients will receive IV lidocaine 1.5 mg/ kg diluted up to 10 ml with normal saline immediately before induction of anesthesia and 10 ml of normal saline infused over 10 min before induction of anesthesia.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive IV dexmedetomidine 0.5 μg /kg diluted up to 10 ml with normal saline infused over 10 min before induction of anesthesia, and 10 ml of normal saline immediately before induction of anesthesia.
  Arms: Group D
Drug: Magnesium sulphate — Patients will receive IV magnesium sulphate 50 mg/kg diluted up to 10 ml with normal saline infused slowly over 10 min before induction of anesthesia, and 10 ml of normal saline immediately before induction of anesthesia.
  Arms: Group M
Drug: Lidocaine — Patients will receive IV lidocaine 1.5 mg/ kg diluted up to 10 ml with normal saline immediately before induction of anesthesia and 10 ml of normal saline infused over 10 min before induction of anesthesia.
  Arms: Group L

SUMMARY:
Laryngoscopy and endotracheal intubation are necessary for effective control of airway and ventilation, but it has deleterious effects such as hypertension and disrhythmia

DETAILED DESCRIPTION:
Fast-track laparoscopic gynecological surgery usually done under general anesthesia (GA). Laryngoscopy and endotracheal intubation are necessary for effective control of airway and ventilation, but it has deleterious effects such as hypertension and disrhythmia. These hemodynamic changes are due to the reflex sympathetic activity and the magnitude of response is directly proportional to the duration and strength of laryngoscopy. Several drugs and techniques have been tried to attenuate the stress response to laryngoscopy and endotracheal intubation, but none of them have proven to be ideal.

Lidocaine is an amide synthetic local anesthetic, which is used in treatment of ventricular dysrhythmias and as a prophylaxis in ventricular tachyarrhythmia. It has cardio stabilizing action.

Bromage showed that its intravenous (IV) use blunted pressure response to intubation. An IV dose of lidocaine 1.5 mg/kg has been proved to attenuate stress responses during laryngoscopy and intubation.

Dexmedetomidine is a highly selective alpha 2 receptor agonist and possesses the properties of sedation, analgesia, and opioid sparing effect. It has been shown to reduce the laryngeal stress response, reduce the requirement of intravenous (IV) anesthetics, and provides hemodynamic stability.

Magnesium sulphate (Mg SO4) is the fourth most abundant cation in the body and the second most abundant intracellular cation. It activates many of the enzyme system. Mg SO4 inhibits the release of catecholamines from the adrenal medulla and adrenergic nerve endings and is effective in attenuating the blood pressure (BP) response to tracheal intubation. Puri et al showed that MgSO4 50 mg/kg administered before laryngoscopy could attenuate the pressor response to tracheal intubation better than lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Age between 23 to 40 years
* With airway of Mallampati grade I and II
* Elective diagnostic laparoscopic gynecologic surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* Mallampatti grading III and IV, anticipated difficult intubation
* Body mass index (BMI > 35 kg/m2), full stomach, pregnancy
* Emergency surgery
* History of cardiac or neurological disease or patient with asthma
* History of Hypersensitivity to the study drugs
* Advanced hepatic or renal failure.
* Patients in whom the duration of laryngoscopy lasted more than 20 seconds
* Patient refusal.

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-01-03 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate (HR) | 10 minutes before intubation to one hour after surgery
  Beats/ minute